CLINICAL TRIAL: NCT03318952
Title: Efficacy of Articaine vs. Lidocaine When Used for Local Infiltration in Pediatric Dental Procedures
Brief Title: Articaine vs Lidocaine for Pediatric Dental Procedures
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The research did not start and the PI transitioned to another institution.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-33755
Record Dates: First submitted 2017-10-05; First posted 2017-10-24 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Anesthesia, Dental; Pain, Postoperative
Keywords: lidocaine injection; articaine injections; pediatric dental anesthesia; post dental procedure pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Anesthetics, Local; Carticaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- lidocaine then articaine (Experimental): For the first dental procedure 2% lidocaine with 1:100,000 epinephrine will be administered with a buccal infiltration injection followed by 2-3 interpapillary injections and possibly more if needed. For the second dental procedure a single buccal infiltration injection of 4% articaine with 1:100,000 epinephrine will be administered.
  Interventions: Drug: lidocaine; Drug: articaine
- articaine then lidocaine (Experimental): For the first dental procedure a single buccal infiltration injection of 4% articaine with 1:100,000 epinephrine will be administered. For the second dental procedure 2% lidocaine with 1:100,000 epinephrine will be administered with a buccal infiltration injection followed by 2-3 interpapillary injections and possibly more if needed.
  Interventions: Drug: lidocaine; Drug: articaine

INTERVENTIONS:
Drug: lidocaine — A buccal infiltration injection followed by 2-3 interpapillary injections and possibly more if needed of 2% lidocaine with 1:100,000 epinephrine will be administered.
  Other Names: local anesthetic
Drug: articaine — A single buccal infiltration injection of 4% articaine with 1:100,000 epinephrine will be administered
  Other Names: local anesthetic

SUMMARY:
The purpose of this study is to compare the efficacy of two types of local anesthesia (articaine and lidocaine) for infiltration anesthesia during restorative dental procedures on lower teeth in pediatric patients. The patients will require similar dental operative procedures on both right and left sides of the mandible in order to qualify for this study. The study will require at least two dental appointments, where a randomized, cross-over study methodology will be utilized. All subjects will be treated by the same dentist. The comfort of the patient will be assessed at various points during the procedure using the Wong-Baker Faces Scale.

DETAILED DESCRIPTION:
This study will compare articaine to lidocaine with overall quality of anesthesia. When administering lidocaine, the investigator will follow standard of care by administering a buccal infiltration injection followed by 2-3 interpapillary injections, one at each gingival papilla where the rubber dam clamp will be placed and possibly more if needed in areas where dental treatment will be provided. A single buccal infiltration injection of articaine will be administered, with the hypothesis that articaine is a stronger anesthestic and will deliver palatal anesthesia with a single injection, eliminating the interpapillary injections required for lidocaine to achieve adequate soft tissue anesthesia. The comfort of the patient during multiple steps of the dental treatment will be recorded. A randomized, cross-over methodology will be used. This study seeks to find whether adequate anesthesia in the mandible can be achieved with a single injection of articaine in the buccal aspect of the jaw instead of having to administer multiple injections of lidocaine, which can increase patient anxiety and discomfort. By decreasing the number of injections needed for children during dental treatment while providing adequate local anesthesia, dentists can provide more comfortable care to their pediatric patients.

Specific Aims/ Hypothesis

-Specific Aim 1: To compare articaine to lidocaine with achieving effective local anesthesia in the mandible and upper arch of pediatric dental patients.

Hypothesis: The solubility of articaine will provide more effective anesthetic delivery through the soft and hard tissue of the mandible following buccal infiltration, eliminating the need for multiple injections.

-Specific Aim 2: To identify which type of anesthetic provides the best patient experience by way of measuring patient comfort at various stages of the dental procedure.

Hypothesis: The patient will have an equally comfortable experience during the dental procedure when articaine or lidocaine is used.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving dental care at Boston Medical Center Pediatric Dental Clinic, Boston University Pediatric Oral Health Center, and East Boston Neighborhood Health Center Pediatric Dental Clinic
* Patients needing similar restorative dental procedures to primary molar teeth on both sides of the maxillary arch or upper arch
* Boys and girls between ages 4 to 14 years
* English speaking and be able to understand verbal assent.

Exclusion Criteria:

* Patients for whom the use of articaine is contraindicated such as patients with Acetylcholine esterase deficiency
* Patients for whom the use of lidocaine is contraindicated in patients taking metronidazole

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Pain during anesthesia injection using the Wong-Baker faces scale | Anesthesia injection is usually about 10 min before the dental procedure starts.
  Wong-Baker faces scale is a set of six cartoon faces with varying facial expressions ranging from a smile/laughter to tears. Each face has a numeric value with a range of 1 to 10. The higher the numeric value the more intense the pain.
Pain during rubber dam placement using the Wong-Baker faces scale | Rubberdam placement is usually about 5 min before the dental procedure starts.
  Wong-Baker faces scale is a set of six cartoon faces with varying facial expressions ranging from a smile/laughter to tears. Each face has a numeric value with a range of 1 to 10. The higher the numeric value the more intense the pain.
Pain during tooth preparation using the Wong-Baker faces scale | Tooth preparation occurs during the dental procedure.
  Wong-Baker faces scale is a set of six cartoon faces with varying facial expressions ranging from a smile/laughter to tears. Each face has a numeric value with a range of 1 to 10. The higher the numeric value the more intense the pain.
Pain during pulp opening using the Wong-Baker faces scale | Pulp opening occurs during the dental procedure.
  Wong-Baker faces scale is a set of six cartoon faces with varying facial expressions ranging from a smile/laughter to tears. Each face has a numeric value with a range of 1 to 10. The higher the numeric value the more intense the pain.
Pain during restoration placement using the Wong-Baker faces scale | Restoration placement is at the end of the dental procedure, approximately 1 hour.
  Wong-Baker faces scale is a set of six cartoon faces with varying facial expressions ranging from a smile/laughter to tears. Each face has a numeric value with a range of 1 to 10. The higher the numeric value the more intense the pain.

SECONDARY OUTCOMES:
Additional injections of local anesthetic at the first visit | At the completion of the first visit, approximately 1 hour.
  The number of extra injections to achieve anesthesia will be documented for each participant.
Additional injections of local anesthetic at the second visit | At the completion of the second visit, approximately 1 hour.
  The number of extra injections to achieve anesthesia will be documented for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Jayapriyaa Shanmugham, BDS MPH DrPH, Principal Investigator — BU Henry M. Goldman School of Dental Medicine
Locations (1):
- BU Henry M. Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related publication. — https://www.ncbi.nlm.nih.gov/pubmed/9188235
- See also: Related publication. — http://glidewelldental.com/education/chairside-dental-magazine/volume-5-issue-4/patients-who-make-a-dentist-most-anxious-about-giving-injections/
- See also: Related publication. — https://www.ncbi.nlm.nih.gov/pubmed/10832257
- See also: Related publication. — https://www.ncbi.nlm.nih.gov/pubmed/11217590
- See also: Related publication. — https://www.ncbi.nlm.nih.gov/pubmed/16759322